CLINICAL TRIAL: NCT05942222
Title: Treatment of Rhinosinusitis With Nasal Polyposis With Dupilumab and Mepolizumab: A Randomized, Multi-centre, Head-to-head Comparison in Real-world Danish Patients
Brief Title: A Real-world, Head-to-head Comparison of Dupilumab Versus Mepolizumab in Danish Patients With Chronic Rhinosinusitis With Nasal Polyps
Acronym: TORNADO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Korsgaard Pedersen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-ENT-3
Record Dates: First submitted 2023-05-22; First posted 2023-07-12 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Asthma; Eosinophilic; Eosinophilia
MeSH Terms: conditions — Pulmonary Eosinophilia; Eosinophilia | interventions — dupilumab; mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dupilumab week 0-24 300 mg/2 weeks (Active Comparator): Normal dose and interval of Dupixent i.e. 300 mg s.c. every 2 weeks
  Interventions: Biological: dupilumab
- Mepolizumab week 0-24 100 mg/4 weeks (Active Comparator): Normal dose and interval of Nucala i.e. 100 mg s.c. every 4 weeks
  Interventions: Biological: mepolizumab
- Dupilumab week 24-48 300 mg/4 weeks (Active Comparator): Increased dosage interval of Dupixent i.e. 300 mg s.c. every 4 weeks - for subjects on Dupixent who met the 24 weeks effect criteria
  Interventions: Biological: dupilumab
- Dupilumab week 24-48 300 mg/2 weeks (Active Comparator): Normal dose and interval of Dupixent i.e. 300 mg s.c. every 2 weeks but for subjects who have crossed over after 24 weeks due to unmet effect criteria.
  Interventions: Biological: dupilumab
- Mepolizumab week 24-48 100 mg/4 weeks (Active Comparator): Normal dose and interval of Nucala i.e. 100 mg s.c. every 4 weeks but for subjects who have crossed-over after 24 weeks due to unmet effect criteria.
  Interventions: Biological: mepolizumab

INTERVENTIONS:
Biological: dupilumab — Subcutaneus injections in standard doses, i.e. 300 mg s.c. every 2 weeks.
  Other Names: Dupixent
  Arms: Dupilumab week 0-24 300 mg/2 weeks; Dupilumab week 24-48 300 mg/2 weeks; Dupilumab week 24-48 300 mg/4 weeks
Biological: mepolizumab — Subcutaneus injections in standard doses, i.e. 100 mg s.c. every 4 weeks.
  Other Names: Nucala
  Arms: Mepolizumab week 0-24 100 mg/4 weeks; Mepolizumab week 24-48 100 mg/4 weeks

SUMMARY:
The goal of this randomized clinical trial is to compare the effects of two newly available biological drugs for the treatment of severe chronic rhinosinusitis with nasal polyps in Danish patients.

The main questions it aims to answer are whether the two drugs are comparable in effect after 24 weeks in terms of:

* A subjective score (the SNOT-22)
* An objective score, i.e.the physician-assessed score of nasal polyp size (the Nasal Polyp Score (0-8))

Methods:

Participants will be randomized to receive one of the IMPs drug in the standard dose. After 24 weeks the effect is assessed by subjective and objective measures. If the criteria set by the Danish Medicinal Council are met (see elsewhere), treatment continues with the same drug for an additional 24 weeks. If the effect criteria are not met, the subject crosses-over to the opposite drug for an additional 24 weeks. After 48 weeks the effect is assessed once more.

DETAILED DESCRIPTION:
Objectives:

* The primary objective is to

  1. establish non-inferiority of dupilumab versus mepolizumab, and if that is established, then
  2. test for possible superiority of dupilumab over mepolizumab in the following hierarchical order (SNOT-22 - Sniffin' Sticks 16 - NPS - ACQ
* The secondary objective is to explore any other relevant differences between mepolizumab and dupilumab in terms of frequency of AEs, need for rescue treatments, diversity in outcome based on endotype or comorbidity or other factors, that can lead to a patient-centred approach, when choosing treatment for CRSwNP.

Trial design:

A randomized, multi-center non-inferiority trial (phase IV RCT). The trial is unblinded.

Investigational medicinal products (IMPs) will be "off-the-shelf" and administered in EMA-approved dosages and -intervals.

Trial population:

The trial aims to include 220 patients with severe, uncontrolled CRSwNP (110 patients in each treatment group). The patients will be recruited from 9 different sites across Denmark. Treatment in Denmark is 100% subsidized by the state.

Methods:

Subjects fulfilling inclusion criteria will be randomized 1:1 to either dupilumab or mepolizumab. After 24 weeks a halfway evaluation will decide if subjects are to stay in their current treatment arm, or cross-over to the opposite arm.

By including 220 participants (effectively 176 participants after 20% drop-outs) the study will achieve a power of >95% to show non-inferiority of dupilumab to mepolizumab for both co-primary endpoints with the following criteria: Level of significance for both endpoints of a one-sided test, p<0.025 and including previously found standard deviation (SD) values 1.9 for NPS and 22 for SNOT-22, an expected superior effect of 0.7 for NPS and 7 on SNOT-22, a minimal clinically relevant difference (MCID) of 1 for NPS and 12 for SNOT-22, respectively.

Trial medication:

All trial medication will be "off the shelf" i.e. no special labelling. It will be provided by hospital pharmacies in accordance with GMP. The investigational medicinal products (IMPs) are dupilumab (Dupixent, Sanofi) and mepolizumab (Nucala, GSK). Dupilumab are administered as subcutaneous injections of 300 mg every two weeks in the first 24 weeks. If the DMC response criteria (table 2) are met after 24 weeks, the dosing interval will be increased to every four weeks, in accordance with previous research and DMC recommendations. Mepolizumab is administered subcutaneously as 100 mg sc. every four weeks. Patients will continue standard of care treatment of INCS and saline irrigation, unless contraindicated.

If rescue treatment is needed, a course of oral corticosteroids (Prednisolone) 37.5 mg once daily for 7 days will be given.

Trial schedule:

Planned first subject first visit May 2023

Planned last subject randomized February 2025

Planned last subject last visit:March 2026

End of trial March 2026

ELIGIBILITY:
Inclusion Criteria:

* Bilateral polyps in nose and sinuses
* ESS within the last three years (unless unfit for surgery y- in this study defined as either a severe somatic disease, for which other specialist advise against surgery, e.g., cardiac disease, pulmonary disease, or coagulation disorder OR/AND severe anxiety which can either be due to previous traumatic experiences with surgery or the postoperative period, post-traumatic stress disorder or severe anxiety disorder. In cases of doubt, investigators can ask for a written statement from the general practitioner or a psychiatrists/psychologist))
* Optimal local treatment with saline irrigation and topical nasal steroids for at least three months (unless contraindicated)
* Evidence of type 2 inflammation

Furthermore, patients must fulfil three out the following five criteria:

* Need for systemic corticosteroids (at least two courses/year OR long-term treatment >3 months) or contraindication to systemic steroids
* Significantly impaired QoL (SNOT-22 score≥50)
* Significant LoS (SSIT-16 score 0-8)
* NPS ≥5 (with at least 2 on either side)
* Asthma diagnosis (requiring inhaled corticosteroid (ICS))

Also: Age of 18 years or more and able to read and/or speak Danish

Exclusion criteria

* Systemic corticosteroid treatment within the last three months
* Endoscopic sinus surgery (ESS) within the last six months
* Non-adherent to medicine regimens
* Hypersensitivity to the active substance or any of the excipients in the two IMPs
* Not able to understand spoken and/or written Danish
* Participation-current or previous (within the last year)-in another investigational drug trial with monoclonal antibodies for asthma, CRSwNP, atopic dermatitis or allergic rhinitis.
* Previous treatment failure with one of the IMPs for any indication (treatment failure is defined as failure to achieve the desired therapeutic outcome or effectively manage a condition within an expected timeframe)
* Eosinophilic blood cell count of ≥1.5x10^9cells/L (at baseline, i.e. before first injection)
* Pronounced fear of needles
* Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
SNOT-22 | Week 24
  Sino-Nasal Outcome Test 22 - change in score since baseline is measured.
NPS | Week 24
  Nasal Polyp Score (0-8): 0 is no polyps, 4 is polyps extending below inferior turbinate's lower border. Each side is scored. The change in score at week 24 since baseline is measured.

SECONDARY OUTCOMES:
SNOT-22 | Week 48
  Sino-Nasal Outcome Test 22 - change in score since week 24 and week 0 if applicable
NPS | Week 48
  Nasal Polyp Score (0-8): 0 is no polyps, 4 is polyps extending below inferior turbinate - lower border. Each side is scored. Change in score since week 24 and week 0 if applicable
Smell score (Sniffin' Sticks Identification Test-16- SSIT-16) | Week 48
  Change since baseline in SSIT-16 (range 0-16, where 0-8 is anosmia)
Asthma control (Asthma Control Questionnaire) | Week 48
  Proportion of patients with ACQ score > 0,5 indicating well-controlled asthma.
Nasal Congestion Score (NCS) | Week 48
  Range 0-3. Change since baseline
Visual Analogue Scale of: smell/asthma/Chronic rhinosinusitis/N-ERD | Week 48
  Change in VAS-score (range 0-10) since baseline
Proportion meeting the evaluation criteria set by the DMC | Week 48
  The DMC criteria is available at medicinraadets website medicinraadet.dk
Fraction of Nitrous Oxide in expired air (FeNO) | Week 48
  A score above 25 indicates eosinophilic inflammation.
Proportion needing rescue treatment | Week 48
  A rescue treatment is defined as systemic oral corticoids or endoscopic sinus surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pedersen, MD, Principal Investigator — Department of ORL, Head and Neck Surgery & Audiology, Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark; Christian von Buchwald, Study Director — Department of ORL, Head and Neck Surgery & Audiology, Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark
Locations (9):
- Denmark (9):
  - Aalborg Universitetssygehus Syd, Aalborg
  - Aarhus Universitetshospital Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Regionshospitalet Gødstrup, Herning
  - Nordsjællands Hospital, Hillerød
  - Sjællands Universitetshospital Køge, Køge
  - Odense Universitetshospital, Odense
  - Sygehus Lillebælt Vejle, Vejle

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT05942222/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT05942222/SAP_001.pdf